CLINICAL TRIAL: NCT06858345
Title: Study of Maternal and Fetal Cardiovascular Function in Hypertensive States of Pregnancy
Acronym: CARDIAC-OAT
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Other Study IDs: CARDIAC-OAT
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- • Duration of gestation in pregnancy complicated by hypertensive state of pregnancy with antihyperte: • Duration of gestation in pregnancy complicated by hypertensive state of pregnancy with antihypertensive therapy guided by hemodynamic phenotypes

SUMMARY:
The pharmacological treatment strategy is then tailored to the underlying hemodynamic phenotype of each patient. That is, rather than applying a one-size-fits-all treatment for all patients, therapy is tailored to the specific characteristics of how the cardiovascular system functions in each patient (e.g., whether the problem is more related to blood volume, vascular resistance, cardiac output, etc.). The goal is to personalize therapy to more effectively treat hypertensive states of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Women with singleton and twin pregnancies complicated by hypertensive states of pregnancy.

Exclusion Criteria:

* Minors under 18 years of age.
* Women with mental disabilities.
* Major congenital fetal anomaly.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant patients undergoing regular hospital follow-up
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Prolongation of at least one week of gestation in pregnancy complicated by hypertensive state of pregnancy with antihypertensive therapy guided by hemodynamic phenotypes | Up to 40 weeks
  Number of weeks of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- HCUVA, El Palmar, Murcia, Spain